CLINICAL TRIAL: NCT04454892
Title: A Study on the Natural History and Clinical Features of Amyotrophic Lateral Sclerosis (ALS) in Mainland China
Brief Title: Natural History and Clinical Features of Amyotrophic Lateral Sclerosis (ALS)
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUTH2019388
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; Epidemiology
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amyotrophic lateral sclerosis patients: Although previous studies have provided reference for the diagnosis and treatment of ALS, the etiology of ALS is still unknown, and the relevant clinical features and natural history of ALS still lack the verification of large samples. Therefore, the research on the natural history of ALS is of great significance to further increase the understanding of ALS and provide new evidence for the diagnosis and treatment of ALS
  Interventions: Other: Amyotrophic lateral sclerosis

INTERVENTIONS:
Other: Amyotrophic lateral sclerosis — AMYOTROPHIC lateral sclerosis (ALS) is a degenerative disorder of motor neurons in the cortex, brainstem and spinal cord1,2. Its cause is unknown and it is uniformly fatal, typically within five years3

SUMMARY:
1. Describe the distribution of ALS in mainland China, to explore the differences in the number of ALS in different times, regions and populations in order to further explore the causes affecting the distribution of ALS;
2. To investigate the cause of ALS in mainland China in the crowd disease development process and the corresponding characteristics change ;
3. To explore the effect of prognosis of ALS;

DETAILED DESCRIPTION:
With the development of supportive measures, the natural history of ALS has changed. Researchers compared the natural history of ALS patients from 1999-2004 and 1984-1998 and found that the median survival time was significantly longer in the former than in the latter (4.32 years vs. 3.22 years) and that the disease progression was slower in the former, even after adjusting for other confounding factors. Although previous studies have provided reference for the diagnosis and treatment of ALS, the etiology of ALS is still unknown, and the relevant clinical features and natural history of ALS still lack the verification of large samples. Therefore, the research on the natural history of ALS is of great significance to further increase the understanding of ALS and provide new evidence for the diagnosis and treatment of ALS.

ELIGIBILITY:
Inclusion Criteria:

- Patients were diagnosed with ALS recruited from all participant clinical centers.The diagnosis of ALS was made using the revised El Escorial criteria for definite, probable, lab-supported, and possible.

Exclusion Criteria:

* Decline to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ALS patients in mainland China.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years to 10 years after recruitment
  Time interval from disease diagnosis to death
Indicators of disease progression | 1 year to 10 years after recruitment
  1) in the diagnosis of disease progression (⊿ FS) = (diagnosis of FRS - R score - when follow-up FRS - R)/diagnosis and follow-up time 2）Weight loss =(weight at diagnosis - weight at follow-up)/time to follow-up 3) BMI decreased = (BMI) at the time of diagnosis of BMI - follow-up/diagnosis and follow-up time 4) FVC decreased = (FVC - during the diagnosis to follow-up FVC)/diagnosis and follow-up time 5) between the above indexes can also be in all follow-up multiple numerical calculation, observing the trend of the change over time

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD.PHD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No